CLINICAL TRIAL: NCT01264653
Title: Study of Intracameral Adrenaline for Pupil Dilation Without Topical Mydriatics in Refractive Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, A-Yong Yu, A-Yong Yu, Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Wenzhou Medical College
Record Dates: First submitted 2010-12-20; First posted 2010-12-22 (Estimated); Last update posted 2012-07-06 (Estimated); Status verified 2012-07

CONDITIONS: Cataract
Keywords: cataract
MeSH Terms: conditions — Cataract | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- experimental group,control group (Experimental): Intraocular adrenalin,topical mydriatics, experimental group: Intervention: Procedure:refractive cataract surgery with Intraocular adrenalin, control group:refractive cataract surgery with topical mydriatics
  Interventions: Drug: adrenalin

INTERVENTIONS:
Drug: adrenalin — adrenalin 0.01%
  Other Names: adrenaline hydrochloride

SUMMARY:
The purpose of this study is to study the safety and efficacy of intracameral adrenaline for pupil dilation without topical mydriatics in refractive cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* male and female
* can read and sign informed consent form；
* Clinical diagnosis of cataract
* Cataract density grade II-III according to the Emery-Little system classification system

Exclusion Criteria:

* sensitivity to adrenalin；
* sensitivity to topical mydriatics；
* any other ocular surgeries；
* iris abnormalities

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pupil size after intracameral adrenaline | 1day
  We would like to evaluate Pupil size dilated with intracameral adrenaline 0.01%

SECONDARY OUTCOMES:
endothelial cell count | 1month
  we would like to evaluate the endothelial cell count 1 month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ayong Yu, Study Director — Wenzhou Medical University
Locations (1):
- Wenzhou Medical College, Wenzhou, Zhejiang, China